CLINICAL TRIAL: NCT03649035
Title: Use of the Eus-guided Cryothermal Ablation in the Multimodality Approach to Patients With Stage III (Locally Advanced and Borderline Resectable) Pancreatic Adenocarcinoma
Brief Title: Eus-guided Cryothermal Ablation in Stage III Pancreatic Adenocarcinoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped for internal decisions
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Principal Investigator, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTP1
Record Dates: First submitted 2018-08-07; First posted 2018-08-28 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Cancer; Pancreas Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: HTP treatment — Elegible patients will undergo HTP treatment, followed by standard of care Chemo therapy and SBRT protocol.

SUMMARY:
Pancreatic cancer represents the 11th most commonly diagnosed cancer in men and 9th in women, being the third leading cause of cancer-related death in the Western countries. Pancreatic cancer has a very poor prognosis and median overall survival is less than 5 months in population-based studies. Approximately 80% of patients with pancreatic cancer present with unresectable disease, which is either due to locally advanced or metastatic disease. About 40% of patients have metastases at the time of diagnosis and in another 30 to 40 % of the patients tumour resection is not feasible because of vascular invasion, or poor general conditions. In resectable patients surgical resection with negative margins (R0) continues to be worldwide considered the only chance to cure, however, this standard treatment is usually reserved to a small number of patients. In patients with locally advanced tumour, neoadjuvant treatment has been proposed in various modalities as a way to decrease size and downstage the tumour leading to a resectable disease. Several phase I - II studies have shown the capability of chemotherapy alone or chemo radiotherapy based regimens to increase the resection rates of these patients and the related median overall survival.

Systemic chemotherapy followed by chemoRT or stereotattic body radiation therapy (SBRT) is an option for selected patients with unresectable disease and good PS who have not developed metastatic disease.

This sequence is especially recommended in cases in which it is highly unlikely that the patient will become resectable (ie, complete encasement of SMA/superior celiac artery). Due to the significant rate of toxicity of the radio therapy (RT) treatment alone or in adjunct to chemotherapy, other local treatments with the goal to downstage the primary tumour with less or no toxicity as compared to RT have been proposed.

Radiofrequency (RF) has been used with success in solid cancers like the hepatocellular carcinoma while cryoablation has been used for breast and renal cancers. RFA has been applied in few clinical trials in human pancreatic cancer either without any imaging guidance or just under intra-operatory ultrasound control during palliative open surgery.

The HybridTherm probe (HTP), (ERBE Elektromedizin GmbH, Tübingen, Germany) combines bipolar RF-ablation with cryogenic induced cooling. A bipolar radiofrequency system creates ablation with less collateral thermal damage than standard monopolar systems but with the trade-off to lose overall efficiency.

In a recent in-vivo study the feasibility of the HTP in patients with unresectable locally advanced pancreatic adenocarcinoma has been shown. HTP has been applied under EUS-guidance to patients who have been already treated by chemotherapy (two lines) and in many cases with the adjunct of RT.

ELIGIBILITY:
Inclusion criteria:

* Only patients with pathologically proven, locally advanced, unresectable pancreatic adenocarcinoma will be selected.
* The criteria for unresectability will be: encasement or thrombosis of one or more large vessels surrounding the pancreas (celiac axis, portal vein, and/or superior mesenteric artery and/or vein, and/or hepatic artery, except the splenic vessels); infiltration of the vessel wall or contact 180° for more than 2 cm length, with initial stricture of the vessel or alteration of the Doppler signal (each patient will undergo thoracic and abdominal-CT with contrast medium to check resectability and detect the absence of distant metastasis).

Esclusion criteria:

* Patients with pancreatic tumors other than pancreatic adenocarcinoma (PDAC)
* Patients with resectable, borderline resectable or metastatic PDAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with feasible EUS-guided Cryothermal Ablation | The day of procedure
  The procedure will be defined as "feasible" if the placement of the probe inside the tumor will be successful and "not feasible" if it will not be possible to place the probe inside the lesion because of difficulties such as hardness of the tumor, stiffness of the GI wall, or interposition of vessels

SECONDARY OUTCOMES:
Progression-free survival | 6 months after the procedure
  To demonstrate the efficacy of the HybridTherm probe in the control of the tumour progression in terms of progression-free survival, measured at 6-month after therapy onset (PFS-6) by MRI. PFS-6 takes in consideration the tumour growth in relation to the volume/size evaluated as a difference between the previous and the current examination.
  In practice, it is the time interval between the enrolment of the patient and the first radiological evidence of tumor progression.
Number of participants with treatment-related adverse events | 30 days after the procedure
  Complications will be recorded and laboratory and radiologic follow-up will be performed to detect them.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided